CLINICAL TRIAL: NCT00447044
Title: Combined Effects of Nutritional and Exercise Countermeasures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Arny A. Ferrando, PhD, UAMS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 72779
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Muscular Atrophy; Muscle Weakness
Keywords: Muscle loss and Maintenance of Muscle function
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness | interventions — Resistance Training; Amino Acids, Essential

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- 2 (Experimental): Subjects drink essential amino acid supplement 3x day for 2 days.
  Interventions: Dietary Supplement: essential amino acids
- 1 (Placebo Comparator): Subjects receive inert substance versus protein supplement.
  Interventions: Dietary Supplement: diet orange soda
- 3 (Experimental): Resistance exercise.
  Interventions: Behavioral: Resistance Exercise

INTERVENTIONS:
Behavioral: Resistance Exercise — Subjects will lift weights with their legs.
  Arms: 3
Dietary Supplement: diet orange soda — Subjects drink diet orange soda 3x day for 2 days.
  Arms: 1
Dietary Supplement: essential amino acids — Subjects drink 15 grams of EAA mixed into diet orange soda 3x day for 2 days.
  Arms: 2

SUMMARY:
The purpose of this study is to see if a combination of resistance exercises and amino acid capsules can reduce muscle loss and maintain muscle function during bedrest. This experiment will imitate many of the physical conditions experienced by astronauts during space flight by examining the effects of resistance exercise or nutrition on muscle during 2 days of bedrest. The diet of astronauts will also be imitated by providing diets in the General Clinic Research Center.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age
* Availability of transport and ability to report to Research Center at appointed times

Exclusion Criteria:

* Subjects with limiting or unstable angina or a cardiology confirmed ECG which demonstrates cardiac abnormalities such as > 0.2 mV horizontal or downsloping ST segment depression, frequent arrhythmia's (>10 PVC/min), or valvular disease.
* Subjects with vascular disease as determined by a combination of risk factors of peripheral atherosclerosis, namely hypertension, obesity, diabetes, hypercholesterolemia and/or evidence of venous or arterial insufficiency upon palpitation of femoral, popliteal, and pedal arteries.
* Any history of hypo- or hyper-coagulation disorders including subjects taking Coumadin or with a history of DVT or PE at any point in their lifetime.
* Any subject that has a chronically elevated systolic pressure >170 or a diastolic blood pressure > 100 will be excluded. Subjects may be included if they are taking blood pressure medication and have a blood pressure below these criteria.
* Any subject with an uncontrolled metabolic disease including liver or renal disease.
* Fasting blood glucose of >126 mg/dl on two separate occasions
* Presence of acute illness or metabolically unstable chronic illness.
* Any subject currently on weight-loss diet.
* Inability to abstain from smoking for duration of study.
* Recent ingestion of anabolic steroids (within 6 months).
* Subjects with atrial fibrillation, history of syncope, angina or congestive heart failure.
* Subjects with a recently (6 months) treated cancer other than Basal Cell Carcinoma.
* Pregnancy/lactation.
* Any other condition or event considered exclusionary by the PI and covering faculty

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Fractional synthetic rate of muscle growth. | two days.

CONTACTS AND LOCATIONS:
Overall Officials: Arny Ferrando, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States